CLINICAL TRIAL: NCT03459248
Title: Metoclopramide-Ondansetron Dual Therapy vs Metoclopramide Monotherapy for Treatment of Nausea and Vomiting Post Laparoscopic Cholecystectomy
Brief Title: Metoclopramide-Ondansetron vs. Metoclopramide Therapy for Treatment of Nausea and Vomiting Post Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 122018
Record Dates: First submitted 2018-03-03; First posted 2018-03-08 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dual Anti-Platelet Therapy; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual therapy (Experimental): Patients will receive 10 mg metoclopramide with 4mg ondansetron before induction of general anesthesia
  Interventions: Other: Dual therapy; Other: General anesthesia
- Monotherapy (Active Comparator): Patients will receive 10 mg metoclopramide before induction of general anesthesia.
  Interventions: Other: Monotherapy; Other: General anesthesia

INTERVENTIONS:
Other: Dual therapy — combination of 10 mg metoclopramide with 4 mg ondansetron
  Arms: Dual therapy
Other: Monotherapy — 10 mg metoclopramide
  Arms: Monotherapy
Other: General anesthesia — Induction of general anesthesia will be performed followed by endotracheal intubation.

SUMMARY:
The incidence of postoperative nausea and vomiting (PONV) after general anesthesia is up to 30% when inhalational anesthetics are used with no prophylaxis. This makes PONV one of the most common complaints following surgery under general anesthesia, together with postoperative pain.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind controlled clinical trial. Written informed consent will be obtained from patients. Patients will be randomly assigned using the sealed envelope technique into 2 equal groups:

Group 1: Patients will receive 10 mg metoclopramide with 4mg ondansetron before induction of general anesthesia.

Group 2: Patients will receive 10 mg metoclopramide before induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging 16 years and above
* Patients undergoing laparoscopic cholecystectomy under General Anesthesia at Makassed General Hospital

Exclusion Criteria:

* Patients with history of motion sickness
* Patients on previous treatment by anti-emetics for dizziness, vertigo or other causes of nausea and vomiting
* Patients with any type of allergy to metoclopramide or ondansetron
* Patients refusing to be part of the study (refusal to sign consent)
* Patients on previous treatment by opioids

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 36 hours postoperatively
  The Primary aim of this study is to compare the effect of prophylactic combination therapy (dual therapy) metoclopramide-ondansetron vs. ondansetron monotherapy for the treatment of postoperative nausea and vomiting after laparoscopic cholecystectomy. This will be assessed through a questionnaire with yes or no question where yes indicates the presence of nausea or vomiting and no indicating the absence of nausea or vomiting.

SECONDARY OUTCOMES:
Surgeon satisfaction | 36 hours postoperatively
  Assess surgeon satisfaction with anesthesia using a questionnaire named "the Surgeon Satisfaction with Anesthesia Services Scales". The questionnaire uses a scale: 1-strongly disagree, 2- disagree, 3- agree, 4- strongly agree
Patient satisfaction | 36 hours postoperatively
  Assess patient satisfaction with anesthesia using the Iowa Satisfaction Anesthesia scale which measures patient satisfaction through a scale: strongly disagree, disagree, undecided, agree and strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon